CLINICAL TRIAL: NCT07369518
Title: Effect of Ceftazidime-Avibactam Against Carbapenemase-Positive Klebsiella Pneumoniae Causing Health Care-Associated Infections
Brief Title: Effect of Ceftazidime-Avibactam on Carbapenemase-Producing Klebsiella Pneumoniae
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Walaa ismail Marzouk, Demonstrator at medical microbiology and immunology department faculty of medicine so, Sohag University
Other Study IDs: Soh-Med-25-12-2MS
Record Dates: First submitted 2026-01-10; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: ISOLATION OF KLEB. by Culture on macConkey Agar; Antibiotic Sensitivity Testing of Different Antibiotics According to Clsi 25; Effect of Ceftazidime-Avibactam on Carbapenemase-Producing Klebsiella Pneumoniae; Detection of Resistance Gene in Isolates Using Conventional Pcr; Detection of Some Virulence Genes Using Conventional Pcr

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 patients with klebsiella pneumoniae infection: Infections caused by klebsiella pneumoniae like skin infections, chest infections, surgical site infections, and urinary tract Infections.
  Interventions: Genetic: . - Genotypic detection of carbapenemase genes by conventional PCR.
- Group 2 patients without klebsiella pneumoniae: Infections caused by any organisms other than klebsiella pneumoniae and carbapenem resistant klebsiella pneumoniae by mechanism other than carbapenemases production.
  Interventions: Genetic: . - Genotypic detection of carbapenemase genes by conventional PCR.

INTERVENTIONS:
Genetic: . - Genotypic detection of carbapenemase genes by conventional PCR. — Specimen Collection : Clinical specimens included blood, urine, bronchoalveolar lavage fluid, wound, peritoneal fluid, and tracheal aspirate obtained from patients with suspected bacterial infections collected in dry sterile well-closed plastic cups. Bacterial identification by Gram stain, culture and biochemical rections - analysisThe resistance pattern of the isolates will be detected by disc diffusion method. - phenotypic detection of carbapenemases. • Detection of carbapenem resistance genes (KPC, VIM, IMP, OXA-48, NDM) by conventional PCR.

SUMMARY:
Specimen Collection : Clinical specimens included blood, urine, bronchoalveolar lavage fluid, wound, peritoneal fluid, and tracheal aspirate obtained from patients with suspected bacterial infections collected in dry sterile well-closed plastic cups.

Bacterial identification by Gram stain, culture and biochemical rections

* analysisThe resistance pattern of the isolates will be detected by disc diffusion method.
* phenotypic detection of carbapenemases. • Detection of carbapenem resistance genes (KPC, VIM, IMP, OXA-48, NDM) by conventional PCR.

DETAILED DESCRIPTION:
Carbapenem-resistant Enterobacterales (CRE) poses an urgent global public health threat, with more than 1,100 documented deaths, as reported in a 2019 antibiotic resistance publication by the U.S. Centers for Disease Control and Prevention.

Carbapenem-resistant Enterobacterales, including carbapenem-resistant Klebsiella pneumoniae (CRKP), is associated with higher mortality compared with infections caused by carbapenem-susceptible Enterobacterales infections Specimen Collection : Clinical specimens included blood, urine, bronchoalveolar lavage fluid, wound, peritoneal fluid, and tracheal aspirate obtained from patients with suspected bacterial infections collected in dry sterile well-closed plastic cups.

Bacterial identification by Gram stain, culture and biochemical rections

* analysisThe resistance pattern of the isolates will be detected by disc diffusion method.
* phenotypic detection of carbapenemases. • Detection of carbapenem resistance genes (KPC, VIM, IMP, OXA-48, NDM) by conventional PCR.

ELIGIBILITY:
Inclusion Criteria: Infections caused by klebsiella pneumoniae like skin infections, chest infections, surgical site infections, and urinary tract Infections.-

Exclusion Criteria:

* Infections caused by any organisms other than klebsiella pneumoniae and carbapenem resistant klebsiella pneumoniae by mechanism other than carbapenemases production.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All selected patients subjected to complete history All samples transported to medical microbiology department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
1 ISOLATION OF KLEB. by culture on macConkey agar | 6 months from January to may
Antibiotic sensitivity testing of different antibiotics according to clsi 25 | 6 months from January to may
Effect of Ceftazidime-Avibactam on Carbapenemase-Producing Klebsiella Pneumoniae | 6 months from January to may
Detection of resistance gene in isolates using conventional pcr | 6 months from June to December
Detection of some virulence genes using conventional pcr | 6 months from June to December

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No